CLINICAL TRIAL: NCT00772629
Title: Antibody Responses Following Meningococcal Tetravalent (A, C, Y, and W-135) Conjugate Vaccination in Healthy Adults Who Were Either Previously Vaccinated With Unconjugated Meningococcal Polysaccharide (Serogroups A, C or Serogroups A, C, Y, and W-135) Vaccine or Not Vaccinated With Meningococcal Vaccine
Brief Title: Antibody Responses Following Meningococcal Tetravalent (A, C, Y, and W-135) Conjugate Vaccination in Healthy Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See detailed description for termination reason
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTA16
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Results first posted 2009-04-27 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-01

CONDITIONS: Meningitis; Meningococcemia
Keywords: Menactra®; Meningitis; Meningococcemia; Neisseria meningitidis
MeSH Terms: conditions — Meningitis; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Subjects naïve to any meningococcal vaccination
  Interventions: Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate
- Group 2 (Experimental): Subjects who previously received unconjugated polysaccharide vaccine (either bivalent A and C or tetravalent A, C, Y, and W 135)
  Interventions: Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate

INTERVENTIONS:
Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Group 1
Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Group 2

SUMMARY:
This study was designed to generate data for the assessment of Meningococcal Polysaccharide Diphtheria Toxoid Conjugate vaccine (Menactra®) when given to adults aged 18 to 55 years.

Primary Objective:

To describe the antibody response to each serogroup prior to, and 4 to 6 weeks following, the administration of one dose of the investigational Meningococcal Polysaccharide Diphtheria Toxoid Conjugate vaccine (Menactra®), as measured by serum bactericidal activity using baby rabbit complement (SBA BR) in participants in each of the two study groups.

Secondary Objective:

To collect reference sera for the development and refinement of laboratory assays for the measurement of antibody responses to serogroups Y and W 135.

DETAILED DESCRIPTION:
Enrollment was terminated before the planned sample size was achieved because the principal investigator and the Sponsor decided that sufficient sera had been obtained to meet the secondary objective of the study.

There were no safety concerns involved in the decision to stop enrollment. Subjects that were enrolled at the time completed the study as per protocol, the last subject last visit was on 29 April 2004.

ELIGIBILITY:
Inclusion Criteria :

* Participant was at least 18 years of age but not yet 56 years of age at the time of vaccination.
* Participant had received either unconjugated meningococcal polysaccharide (serogroups A and C, or A, C, Y, and W 135) vaccine at least one year prior to enrollment (for assignment to Group 2) or had no prior history of meningococcal vaccination (for assignment to Group 1).
* Participant had signed Ethics Committee-approved informed consent form.

Exclusion Criteria :

* Serious chronic disease (i.e., cardiac, renal, neurologic, metabolic, rheumatologic, psychiatric, etc.)
* Known or suspected impairment of immunologic function
* Acute medical illness with or without fever within the last 72 hours or an oral temperature ≥ 38°C at the time of inclusion
* History of documented invasive meningococcal disease
* Administration of immune globulin or other blood products within the last three months, or injected or oral corticosteroids or other immunomodulatory therapy within six weeks of the study vaccine. Individuals on a tapering dose schedule of oral steroids lasting < 7 days were allowed to be included in the trial as long as they had not received more than one course within the last two weeks prior to enrollment.
* Antibiotic therapy within the 72 hours prior to vaccination or 72 hours prior to drawing the blood sample at Visit 2
* Received unconjugated meningococcal polysaccharide (serogroups A and C, or A, C, Y, and W 135) vaccine within the one-year period prior to enrollment or a conjugated meningococcal vaccine at any time prior to enrollment
* Received any vaccine in the 28-day period prior to enrollment, or scheduled to receive any vaccination during participation in the study
* Suspected or known hypersensitivity to any of the vaccine components
* Unavailable for the entire study period, or unable to attend the scheduled visits or to comply with the study procedures
* Enrolled in another clinical trial
* In females, pregnancy confirmed by positive urine test result
* In females, current breastfeeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2004-01; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (2):
- United Kingdom (2):
  - Bristol
  - London

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 26 January to 29 April 2004 at 2 Medical clinics in the United Kingdom
Pre-assignment Details: Eighteen (18) participants that met the inclusion and exclusion criteria were enrolled. One whom no baseline blood sample could be obtained at Visit 1 was not vaccinated and withdrew from the study.
Groups:
- Meningococcal Vaccine-naive Group: Participants have never received any meningococcal vaccine in the past
- Meningococcal Vaccine-primed Group: Participants who previously received unconjugated polysaccharide vaccine (either bivalent A and C or tetravalent A, C, Y, and W 135
Period: Overall Study
Arm/Group | Meningococcal Vaccine-naive Group | Meningococcal Vaccine-primed Group
Started | 17 | 1
Completed | 16 | 1
Not Completed | 1 | 0
Not completed — Subject was not vaccinated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Meningococcal Vaccine-naive Group | Meningococcal Vaccine-primed Group | Total
Number analyzed (Participants) | 17 | 1 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 1 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.8 (10.20) | 43.0 (0) | 36.2 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 0 | 13
  Male | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United Kingdom | 17 | 1 | 18

OUTCOME MEASURES:

1. Primary Outcome: Participants With a ≥ 4-fold Rise in Antibody Titers as Measured by Serum Bactericidal Assay (SBA) From Day 0 to Day 28.
Description: Number of participants with a minimum of 4 fold rise in Antibody Titers as Measured SBA to each vaccine meningococcal serogroups from Baseline to Day 28.
Time Frame: Day 28 post-vaccination
Population: SBA-BR to each of the 4 meningococcal serogroups in the vaccine was evaluated in the per-protocol population.
Measure: Number; unit: Participants
Arm/Group | Meningococcal Vaccine-naive Group | Meningococcal Vaccine-primed Group
Number analyzed (Participants) | 16 | 1
Participants
  Meningococcal serogroup A | 14 | 0
  Meningococcal serogroup C | 11 | 0
  Meningococcal serogroup Y | 14 | 1
  Meningococcal serogroup W-135 | 15 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination for 42 days post-vaccination.
Arm/Group | Meningococcal Vaccine-naive Group | Meningococcal Vaccine-primed Group
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/1
Other Adverse Events (participants affected / at risk) | 8/16 | 0/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Meningococcal Vaccine-naive Group (N=16) | Meningococcal Vaccine-primed Group (N=1)
Chest pain (General disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 1 | 0
Upper respiratory tract infection NOS (Infections and infestations) | 1 | 0
Viral infection NOS (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Asthma NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Paronychia (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Enrollment was terminated before the planned sample size was achieved because the principal investigator and the Sponsor decided that sufficient sera had been obtained to meet the secondary objective of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.